CLINICAL TRIAL: NCT00886054
Title: The Prediction of Intracranial Pressure and Clinical Outcome by Transcranial Doppler in Neurocritical Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Tsai, Yi-Hsin, Department of Traumatology, National Taiwan University Hospital
Other Study IDs: 200901010R; 97WFA0102463
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Head Injury; Intracerebral Hemorrhage; Ischemic Stroke; Subarachnoid Hemorrhage; Brain Tumor; Hydrocephalus
Keywords: Transcranial Doppler; Transcranial color-coded duplex sonography; Neurocritical patients
MeSH Terms: conditions — Craniocerebral Trauma; Cerebral Hemorrhage; Ischemic Stroke; Subarachnoid Hemorrhage; Brain Neoplasms; Hydrocephalus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Neurocritical patients: Neurocritical patients including those sustaining head injury, cerebrovascular events (such as intracerebral hemorrhage, subarachnoid hemorrhage, etc.), brain tumor, or hydrocephalus.

SUMMARY:
The purpose of this study is to use transcranial Doppler (TCD) to predict intracranial pressure (ICP) and clinical outcome of neurocritical patients.

DETAILED DESCRIPTION:
Transcranial Doppler (TCD) and Transcranial color-coded duplex sonography (TCCS) play an important part in neurocritical monitoring systems. Currently there are studies using flow velocities and pulsatility index (PI) to predict intracranial pressure (ICP) and clinical outcome. But the use of B-mode in such prediction is not yet investigated. The purposes of this study are to establish the correlation among clinical data, CT findings and information collected by TCCS, and to predict ICP and neurological outcome using such information. The focus would be on 3rd ventricle size, midline shift and anteroposterior-transverse ration of midbrain (midbrain index) obtained by B-mode of TCCS. This study is a prospective clinical study targeting on 30 neurocritical patients admitted to intensive care units in one year. The timing of performance of TCCS will be (1) within 6 hours after admission, (2) within 6 hours after each CT examination, and (3) when ICP is higher than 20 mmHg for more than 5 minutes. Glasgow coma scale (GCS), heart rate, blood pressure (systolic, diastolic, and mean), body temperature, central venous pressure (CVP), brain temperature, ICP, cerebral perfusion pressure (CPP), mean velocity (MV) of bilateral middle cerebral arteries (MCAs), PI, midline shift, 3rd ventricular dimension, anteroposterior to transverse ratio of midbrain (midbrain index, MI) are recorded. The latter three parameters are also obtained from CT scans, and compared with those obtained from TCCS. Outcome is evaluated with extended Glasgow outcome scale (GOSE), and analyzed with previous records. This study is going to prove that TCCS is a safe, convenient, real-time and cheap tool in clinical care for neurocritical patients. It also provides prediction of ICP and clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16 to 80 years
* Neurocritical patient (head injury, hemorrhagic or ischemic stroke, subarachnoid hemorrhage, etc.) who was admitted to intensive care unit and had undergone intracranial pressure monitoring

Exclusion Criteria:

* associated with multiple organ impairment or failure
* single organ failure prior to neurocritical condition, such as cardiac, hepatic, or renal failure
* associated with severe infection or sepsis

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted via emergency room for neurosurgical emergency, such as trauma, stroke, etc.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Hsin Tsai, M.D., Principal Investigator — Department of Traumatology, National Taiwan University Hospital
Locations (1):
- Department of Traumatology, National Taiwain University Hospital, Taipei, Taipei, Taiwan

REFERENCES:
- [Background] Aaslid R, Markwalder TM, Nornes H. Noninvasive transcranial Doppler ultrasound recording of flow velocity in basal cerebral arteries. J Neurosurg. 1982 Dec;57(6):769-74. doi: 10.3171/jns.1982.57.6.0769. PMID 7143059
- [Background] Berland LL, Bryan CR, Sekar BC, Moss CN. Sonographic examination of the adult brain. J Clin Ultrasound. 1988 Jun;16(5):337-45. doi: 10.1002/jcu.1870160508. PMID 3152391
- [Background] Bogdahn U, Becker G, Winkler J, Greiner K, Perez J, Meurers B. Transcranial color-coded real-time sonography in adults. Stroke. 1990 Dec;21(12):1680-8. doi: 10.1161/01.str.21.12.1680. PMID 2264074
- [Background] Bor-Seng-Shu E, Hirsch R, Teixeira MJ, De Andrade AF, Marino R Jr. Cerebral hemodynamic changes gauged by transcranial Doppler ultrasonography in patients with posttraumatic brain swelling treated by surgical decompression. J Neurosurg. 2006 Jan;104(1):93-100. doi: 10.3171/jns.2006.104.1.93. PMID 16509152
- [Background] Baussart B, Cheisson G, Compain M, Leblanc PE, Tadie M, Benhamou D, Duranteau J. Multimodal cerebral monitoring and decompressive surgery for the treatment of severe bacterial meningitis with increased intracranial pressure. Acta Anaesthesiol Scand. 2006 Jul;50(6):762-5. doi: 10.1111/j.1399-6576.2006.01038.x. PMID 16987375
- [Background] Mitchell P, Gregson BA, Vindlacheruvu RR, Mendelow AD. Surgical options in ICH including decompressive craniectomy. J Neurol Sci. 2007 Oct 15;261(1-2):89-98. doi: 10.1016/j.jns.2007.04.040. Epub 2007 Jun 4. PMID 17543995
- [Background] Vahedi K, Vicaut E, Mateo J, Kurtz A, Orabi M, Guichard JP, Boutron C, Couvreur G, Rouanet F, Touze E, Guillon B, Carpentier A, Yelnik A, George B, Payen D, Bousser MG; DECIMAL Investigators. Sequential-design, multicenter, randomized, controlled trial of early decompressive craniectomy in malignant middle cerebral artery infarction (DECIMAL Trial). Stroke. 2007 Sep;38(9):2506-17. doi: 10.1161/STROKEAHA.107.485235. Epub 2007 Aug 9. PMID 17690311
- [Background] Tang SC, Huang SJ, Jeng JS, Yip PK. Third ventricle midline shift due to spontaneous supratentorial intracerebral hemorrhage evaluated by transcranial color-coded sonography. J Ultrasound Med. 2006 Feb;25(2):203-9. doi: 10.7863/jum.2006.25.2.203. PMID 16439783
- [Background] Schmidt B, Klingelhofer J, Schwarze JJ, Sander D, Wittich I. Noninvasive prediction of intracranial pressure curves using transcranial Doppler ultrasonography and blood pressure curves. Stroke. 1997 Dec;28(12):2465-72. doi: 10.1161/01.str.28.12.2465. PMID 9412634
- [Background] McQuire JC, Sutcliffe JC, Coats TJ. Early changes in middle cerebral artery blood flow velocity after head injury. J Neurosurg. 1998 Oct;89(4):526-32. doi: 10.3171/jns.1998.89.4.0526. PMID 9761044
- [Background] Newell DW, Aaslid R, Stooss R, Seiler RW, Reulen HJ. Evaluation of hemodynamic responses in head injury patients with transcranial Doppler monitoring. Acta Neurochir (Wien). 1997;139(9):804-17. doi: 10.1007/BF01411398. PMID 9351985
- [Background] Shiogai T, Sato E, Tokitsu M, Hara M, Takeuchi K. Transcranial Doppler monitoring in severe brain damage: relationships between intracranial haemodynamics, brain dysfunction and outcome. Neurol Res. 1990 Dec;12(4):205-13. doi: 10.1080/01616412.1990.11739944. PMID 1982161
- [Background] Marti-Fabregas J, Belvis R, Guardia E, Cocho D, Munoz J, Marruecos L, Marti-Vilalta JL. Prognostic value of Pulsatility Index in acute intracerebral hemorrhage. Neurology. 2003 Oct 28;61(8):1051-6. doi: 10.1212/01.wnl.0000090520.67254.14. PMID 14581663
- [Background] Bouma GJ, Muizelaar JP. Cerebral blood flow in severe clinical head injury. New Horiz. 1995 Aug;3(3):384-94. PMID 7496746
- [Background] Manno EM. Transcranial Doppler ultrasonography in the neurocritical care unit. Crit Care Clin. 1997 Jan;13(1):79-104. doi: 10.1016/s0749-0704(05)70297-9. PMID 9012577
- [Background] Lindegaard KF, Nornes H, Bakke SJ, Sorteberg W, Nakstad P. Cerebral vasospasm diagnosis by means of angiography and blood velocity measurements. Acta Neurochir (Wien). 1989;100(1-2):12-24. doi: 10.1007/BF01405268. PMID 2683600
- [Background] Hunt WE, Hess RM. Surgical risk as related to time of intervention in the repair of intracranial aneurysms. J Neurosurg. 1968 Jan;28(1):14-20. doi: 10.3171/jns.1968.28.1.0014. No abstract available. PMID 5635959
- [Background] Klingelhofer J, Dander D, Holzgraefe M, Bischoff C, Conrad B. Cerebral vasospasm evaluated by transcranial Doppler ultrasonography at different intracranial pressures. J Neurosurg. 1991 Nov;75(5):752-8. doi: 10.3171/jns.1991.75.5.0752. PMID 1919698
- [Background] Wozniak MA, Sloan MA, Rothman MI, Burch CM, Rigamonti D, Permutt T, Numaguchi Y. Detection of vasospasm by transcranial Doppler sonography. The challenges of the anterior and posterior cerebral arteries. J Neuroimaging. 1996 Apr;6(2):87-93. doi: 10.1111/jon19966287. PMID 8634493
- [Result] McCartney JP, Thomas-Lukes KM, Gomez CR. Introduction to Transcranial Doppler. In: Handbook of transcranial Doppler. New York: Springer-Verlag, 1997;1-13.
- [Result] Baumgartner RW. Transcranial color-coded duplex sonography. J Neurol. 1999 Aug;246(8):637-47. doi: 10.1007/s004150050424. PMID 10460438
- [Result] Lindegaard K-F. Indices of pulsatility. In: Newell DW, Aaslid RA, eds. Transcranial Doppler. New York: Raven Press, 1992:67-82.